CLINICAL TRIAL: NCT06840249
Title: Outcomes of Pediatric Vascular Trauma in Assiut University Hospital Trauma Unit
Brief Title: Pediatric Vascular Trauma
Status: Recruiting | Type: Observational
Sponsor: Ahmed Momen Soliman Mohamed (Other)
Responsible Party: Sponsor-Investigator, Ahmed Momen Soliman Mohamed, Assiut University,71515Assiut,Egypt., Assiut University
Organization: Assiut University (Other)
Other Study IDs: Pediatric vascular trauma
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Vascular Trauma
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intervention either by interposition graft or end to end anastomosis or thrombectomy: if vessel injured and no signals intervention is required
  Interventions: Procedure: surgery
- observetional: if patients had good signals no intervention is required

INTERVENTIONS:
Procedure: surgery — surgery by graft or repair or thrombectomy and completion angiography
  Groups: intervention either by interposition graft or end to end anastomosis or thrombectomy

SUMMARY:
pediatric vascular trauma

DETAILED DESCRIPTION:
outcomes of treatment and also observation

ELIGIBILITY:
Inclusion Criteria:

* less than 18 years and more 3yrs

Exclusion Criteria:

* iatrogenic injury in non trauma setting

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All pediatric vascular trauma from age 3 yrs uo to 18 yrs
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
limb salvage rates | Baseline
  0utcomes of treatment modalities of pediatric vascular injury

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Morao S, Ferreira RS, Camacho N, Vital VP, Pascoal J, Ferreira ME, Capitao LM, Goncalves FB. Vascular Trauma in Children-Review from a Major Paediatric Center. Ann Vasc Surg. 2018 May;49:229-233. doi: 10.1016/j.avsg.2017.10.036. Epub 2018 Feb 9. PMID 29428539